CLINICAL TRIAL: NCT03895008
Title: Comparing the Stage-for-Stage Prognosis of Patients With Cardia and Non-cardia Gastric Cancer After Operation.
Brief Title: Comparing the Prognosis of Patients With Cardia and Non-cardia Gastric Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Collaborators: Qinghai People's Hospital (Other); LanZhou University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Other Study IDs: AHQU-2019001
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-03

CONDITIONS: Gastric Cancer
Keywords: Cardia gastric cancer; Non-cardia gastric cancer; Resection; Prognosis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardia gastric cancer: Cardiac gastric cancer is defined as a cancer center lies arising 2-5 cm from the gastric mucosa distal to the esophagogastric junction.
  Interventions: Other: Cardia and Non-cardia gastric cancer
- Non-cardia gastric cancer: Non-cardia gastric cancer is defined as tumors originated from the gastric mucosa distal to the cardia.
  Interventions: Other: Cardia and Non-cardia gastric cancer

INTERVENTIONS:
Other: Cardia and Non-cardia gastric cancer — We classify gastric cancer into cardia gastric cancer and non-cardia gastric cancer.

SUMMARY:
To comparing the stage-for-stage prognosis of patients with cardia and non-cardia gastric cancer after operation.

DETAILED DESCRIPTION:
The aim of this study is to compare the stage-for-stage prognosis of patients with cardia and non-cardia gastric cancer after operation.In this study, patients with cardiac and non-cardiac gastric cancer who undergo radical resection from January 2019 to December 2024 will be included. We will follow up the patient's progression, recurrence time and survival time.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology or cytopathology proven cardia or non-cardia gastric cancer;
2. Operable gastric cancer patients: primary lesions can be completely excision, no distant metastasis;
3. Life expectancy of at least 6 months;
4. ECOG（Eastern Cooperative Oncology Group ） score 0-1;
5. Age: 18~80 years old;
6. Normal hemodynamic indices before the recruitment (including blood cell count and liver/kidney function).

   For example: WBC（White blood cell count ）>4.0×109/L; NEU（Neutrophils）>1.5×109/L; PLT（Platelet）>100×109/L;
7. Roughly normal cardiopulmonary function: No coronary heart disease, myocardial infarction, pulmonary heart disease, refractory hypertension;
8. Not concomitant with other uncontrollable benign diseases before the recruitment;
9. Voluntarily signed the informed consent.

Exclusion Criteria:

1. Advanced gastric cancer patients with distant metastasis and inoperable ;
2. Pregnant or lactating women;
3. Patients who have no desire to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gastric cancer
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-07-08 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival（DFS） | 5 years
  The time from the primary operation to disease recurrence or death.

SECONDARY OUTCOMES:
Overall survival(OS) | 5 years
  OS is defined as the time from the end of radical surgery to death for any reason or at the last follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - People's Hospital of Qinghai Province, Xining, Qinghai

IPD SHARING:
Plan to Share IPD: No